CLINICAL TRIAL: NCT06221176
Title: Translational Biomarkers and Therapeutic Development for Very Young Children Diagnosed with Autism Spectrum Disorder and Co-occurring Anxiety
Brief Title: Biomarkers Research in Anxiety for Validation and Efficacy
Acronym: BRAVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Susan Faja, Associate Professor, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: P00046792
Record Dates: First submitted 2024-01-02; First posted 2024-01-24 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Autism; Autism Spectrum Disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Experimental): Being Brave
  Interventions: Behavioral: Being Brave

INTERVENTIONS:
Behavioral: Being Brave — Being Brave is a manualized cognitive-behavioral (CBT) intervention and includes several features that are well-aligned with the needs of autistic children: (1) an intensive parent component; (2) use of visual aids to lay out coping plans and exposure hierarchies, psychoeducation about recognizing fear and anxiety, and scripted language for coping; (3) repeated practice of well-rehearsed coping plans for novel or challenging situations; and (4) exposure exercises for social anxiety and practice of basic social skills. The intervention includes 16 weekly sessions (1 hour each). Delivery of Being Brave is flexible to allow for additional or less practice or exposure opportunities.

SUMMARY:
A within-subjects design will be used for this preliminary investigation of four biomarkers across two contexts of use: prediction of treatment response (i.e., stratification) and quantification of response (i.e., change).

DETAILED DESCRIPTION:
A within-subjects design will be used for this preliminary investigation of four biomarkers across two contexts of use: prediction of treatment response (i.e., stratification) and quantification of response (i.e., change).

The main questions the study aims to answer are:

* To evaluate the stability of each potential biomarker over a 3-4-week retest period. The biomarkers are hypothesized to have adequate stability (ICC: > .5) in the absence of intervention.
* To determine which baseline biomarker scores predict response to a manualized cognitive behavioral therapy (CBT) program for treating anxiety, Being Brave.
* To determine which biomarkers are sensitive to treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3;0 and 6;11 years old
* A diagnosis of autism spectrum disorder using DSM-5 diagnostic criteria
* A diagnosis of anxiety disorder using DSM-5 diagnostic criteria
* Use of fluent 2-3 word phrases or fluent speech (i.e., Module 2 or 3 for ADOS-2)
* Cognitive ability (either verbal or non-verbal IQ) > 80 using the DAS-2
* A parent/guardian who is willing/able to participate and respond to interviews/surveys in English and willing/able to participate in Being Brave parent training in English and support homework activities.

Exclusion Criteria:

* Presence of seizures
* Premature birth (<36 weeks) or low birth weight (<2500 gms)
* Known genetic or medical disorders (e.g., Fragile X), or injuries (e.g., stroke) with implications for the nervous system or that require regular psychoactive medication that alter EEG/RSA/EDR signal (e.g., anti-convulsants)
* Significant sensory or motor impairment (e.g., blindness)
* Major physical abnormalities
* Exposure to environmental factors that could contribute to neurocognitive delays (significant alcohol exposure in utero, extreme environmental deprivation)
* Previous CBT for anxiety
* Presence of conduct or oppositional defiant disorder or ADHD so severe as to interfere with the child's ability to take part in treatment
* Presence of a primary presenting problem for which the intervention would be inappropriate (e.g., obsessive-compulsive disorder, severe mood disorder, suicidality)
* Psychotic symptoms in the child or parents
* Parent/caregiver who is not fluent in English or English is spoken in the home less than half of the time.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Spence Preschool Anxiety Scale (SPAS) or Spence Anxiety Scale (SCAS) Parent Report | At baseline enrollment visit and post intervention approximately 20 weeks later
  Parents of children ages 3 to 5 will complete the SPAS and parents of 6 year old children will complete the SCAS. These are questionnaires designed to assess the severity of anxiety symptoms in preschool-aged and school-aged children. Scores range from 0-136 with higher scores indicating greater anxiety.

SECONDARY OUTCOMES:
Behavior Assessment System for Children (BASC-3) | At baseline enrollment visit and post intervention approximately 20 weeks later
  The BASC-3 measures adaptive and problem behaviors in the community and home setting. It has a strong foundation in theory and research. Scores range from 20-120 with higher scores indicating greater anxiety.
Pediatric Anxiety Rating Scale (PARS) | At baseline enrollment visit and post intervention approximately 20 weeks later
  The PARS is a checklist which the independent evaluating clinician completes based upon parent interview. The measure is designed to assess the severity of anxiety symptoms associated with social phobia, separation anxiety disorder, and generalized anxiety disorder. Scores range from 0-25 with higher scores indicating greater anxiety.
Clinical Global Impression of Anxiety (CGI-A) Interview | At baseline enrollment visit and post intervention approximately 20 weeks later
  The CGI-A assesses severity and improvement of anxiety using a 7-point Likert scale (from "very much better" to "very much worse"). Based on information collected from the KSADSE, PARS, and Spence, the clinician will rate the global severity of the child's global anxiety and of each individual anxiety disorder. Scores range from 0-8 with higher scores indicating greater anxiety.

OTHER OUTCOMES:
Coping Questionnaire (CQ) | At baseline enrollment visit and post intervention approximately 20 weeks later
  To assess changes in a child's ability to manage specific anxiety-provoking situations, parents rate up to six specific anxiety-provoking situations for their child. Scores range from 6-42 with lower scores indicating lower ability to cope with anxiety.
Family Life Impairment Scale (FLIS) | At baseline enrollment visit and post intervention approximately 20 weeks later
  To assess the extent to which child behavior limits participation in activities typical of families with young children, parents will complete this measure. Scores range from 0-38 with higher scores indicating greater impact of child behavior on family functioning.
Resting EEG Alpha Asymmetry | At baseline, 3-4 weeks later, and at post (approximately 20 weeks later)
  Continuous EEG will be collected while children watch non-social videos for a 4 minute baseline period and again after a brief challenge task (working memory, conversation about feelings). The dependent variable will be EEG alpha power asymmetry (i.e., difference in alpha power between the left and right frontal recording sites)
Late Positive Potential mean Event-related Potentials (ERPs) Amplitude | At baseline, 3-4 weeks later, and at post (approximately 20 weeks later)
  ERPs will be collected while children view digitized and standardized photos of neutral, fearful, angry, and happy expressions (50 per condition). Each trial will consist of a 100ms baseline, 500ms face stimulus, 1200ms post-stimulus period, and variable inter-trial interval of 500-1000ms. The dependent variable will be the ERP mean amplitude at the late positive potential measured between 700-1200ms over anterior leads.
Mean Electrodermal Response (EDR) Amplitude | At baseline, 3-4 weeks later, and at post (approximately 20 weeks later)
  EDR will be collected during a task includes acquisition trials that pair a conditioned stimulus (CS+; a geometric shape) with an aversive tone (i.e., unconditioned stimulus). The second conditioned stimulus (CS-; a different geometric shape) is presented alone. The CS+ and CS- are counterbalanced across children and will be unique at each time point. The Pavlovian Conditioning and Extinction Task will be conducted to measure the rate of EDR habituation during the extinction period. In addition, EDR levels will be explored during a series of challenges in different domains paired with non-challenging tasks that control for the psychomotor demands of the challenge task.
Respiratory sinus arrhythmia (RSA) reactivity | At baseline, 3-4 weeks later, and at post (approximately 20 weeks later)
  RSA will be collected during a validated protocol for assessing autonomic nervous system reactivity in children ages 3 to 6. The protocol includes a series of challenges in different domains paired with non-challenging tasks that control for the psychomotor demands of the challenge task. RSA will also be explored during the extinction period of a conditioning task.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Two Brookline Place, Brookline, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No